CLINICAL TRIAL: NCT07354009
Title: Evaluation of the Efficacy and Safety of iStent in Reducing Intraocular Pressure in Adult Patients With Open-angle Glaucoma and Cataract
Brief Title: Efficacy and Safety of iStent in Reducing Intraocular Pressure in Open-angle Glaucoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-1421
Record Dates: First submitted 2025-11-17; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-10

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PHACO+PC-IOL+iStent (Experimental): Cataract extraction combined with intraocular lens implantation + istent imp
  Interventions: Procedure: PHACO+PC-IOL+iStent
- PHACO+PC-IOL (Sham Comparator): Cataract extraction combined with intraocular lens implantation
  Interventions: Procedure: PHACO+PC-IOL

INTERVENTIONS:
Procedure: PHACO+PC-IOL+iStent — PHACO+PC-IOL+iStent
  Other Names: PHACO+PC-IOL
  Arms: PHACO+PC-IOL+iStent
Procedure: PHACO+PC-IOL — PHACO+PC-IOL
  Arms: PHACO+PC-IOL

SUMMARY:
To evaluate the efficacy and safety of istent inject W in reducing intraocular pressure in Chinese adult patients with open-angle glaucoma complicated with cataract.

DETAILED DESCRIPTION:
Group A: Cataract extraction combined with intraocular lens implantation and iStent implantation; Group B: Cataract extraction combined with intraocular lens implantation. The Intraocular pressure changes at 1 day, 1 week, 1 month, 3 months, 6 months and 12 months were observed and compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Gender is not limited. Applicants must be 18 years old or above;
* Study patients whose eyes were diagnosed with open-angle glaucoma;
* The study eye was diagnosed with cataract and met the conditions for phacoemulsification, with the best corrected visual acuity ≤0.7(patients with the best corrected visual acuity >0.7 who were determined by the researcher to need cataract surgery could be enrolled);
* Angular endoscopy confirmed that the opening Angle of the study eye was normal (defined as Shaffer grade ≥3, and there was no peripheral anterior iris adhesion, polycythemia or other abnormal conditions that might affect the correct placement of the stent);
* The patient is capable and willing to provide written informed consent and participate in the regular postoperative follow-up as required.

Exclusion Criteria:

* Patients with angle-closure, pigmentary or pseudo-exfoliative glaucoma;
* Patients with traumatic, malignant uveitis, neovascular or glaucoma related to vascular diseases;
* Suffering from severe diabetic retinopathy, retinal detachment, central retinal vein or artery occlusion, retinal chromosomal degeneration, macular degeneration, macular edema, and determined by researchers to potentially affect surgical safety;
* Patients with identifiable congenital abnormalities of the anterior chamber Angle;
* Having clinically significant corneal dystrophy, active inflammation or having undergone surgery that may interfere with the reliability of intraocular pressure measurement;
* Patients with retrobulbar tumors, thyroid eye disease, cavernous sinus fistula, Sturge-Weber syndrome or any other disease that may cause elevated venous pressure in the outer sclera;
* Suffering from eye or systemic diseases that affect surgical safety or subsequent examinations;
* Pregnant women, lactating women, women of childbearing age who plan to get pregnant during the research period or are unable to take effective contraceptive measures;
* Failure to follow the doctor's advice;
* Other circumstances where the researcher determines that the patient is not suitable for inclusion

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-07 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
intraocular pressure | Baseline, 1 day, 1 week, 1 month, 3 months, 6 months and 12 months
  intraocular pressure

CONTACTS AND LOCATIONS:
Overall Officials: Kaijun Wang, Study Director — Eye Center, the 2nd Affiliated Hospital, Medical College of Zhejiang Universit
Locations (1):
- Eye Center, the 2nd Affiliated Hospital, Medical College of Zhejiang University, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No